CLINICAL TRIAL: NCT02208713
Title: Intramuscular Transplantation of Autologous Muscle Derived Stem Cell(MDSC) and Adipose Derived Mesenchymal Stem Cells (AD-MSC) in Patients With Facioscapulohumeral Dystrophy (FSHD), Phase I Clinical Trial
Brief Title: Intramuscular Transplantation of Muscle Derived Stem Cell and Adipose Derived Mesenchymal Stem Cells in Patients With Facioscapulohumeral Dystrophy (FSHD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Nerve-007
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Dystrophy
Keywords: FSHD muscle derived stem cell adipose derived mesenchymal stem cell intramuscular injection
MeSH Terms: interventions — Injections, Intramuscular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem cell recipient (Experimental): The patients with FSHD who underwent muscle derived stem cell and Adipose derived mesenchymal stem cell with intramuscular injection.
  Interventions: Biological: Intramuscular injection

INTERVENTIONS:
Biological: Intramuscular injection — Intramuscular injection of stem cells in patients with FSHD.
  Other Names: Intramuscular cell transplantation

SUMMARY:
Facioscapulohumeral Dystrophy is a Autosomal dominant inherited dystrophy with the prevalence of 1:20,000 and it is the third most common dystrophy after the dystrophinopathies and myotonic dystrophy. The symptoms including: Pain, facial weakness, scapular fixator, humeral, truncal, pelvic girdle and lower-extremity weakness, High frequency hearing loss, Retinal telangiectasia . The existing treatments are not effective so, cell therapy is a new hope to improve patients' quality of life. Therefore, We design this clinical trial to evaluate the safety and feasibility of stem cell transplantation.

DETAILED DESCRIPTION:
In this study, we select 15 patients with FSHD based on eligibility criteria. All the patients underwent physical examination, laboratory evaluations, EMG-NCV, muscle sonography and muscle MRI. Then, a sample of patient's muscle is taken from Biceps Femoralis to isolate and culture of MDSC. The AD-MSC is prepared from Royan Adipose Tissue Bank. The patient is admitted in general hospital, and the cell suspensions are injected into biceps, triceps and trapezoids muscles by neurologists. After transplantation, the patients will be under observation for 5 hours and will be discharged if no side effect happen. All the patients will be followed at 1,2,4,6 and 12 months after cell injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-50
2. Both gender
3. Weakness of face muscle
4. FSHD phenotype positive
5. Genetic Test confirmation for FSHD

Exclusion Criteria:

1. Co - morbidities: Heart & respiratory diseases,malignancy, rheumatologic disorders
2. Progressive form of disease
3. Not able to sign the consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Myalsia | 1month
  Evaluation the presence of myalsia 1month after cell injection.
Mass formation | 6 months
  Evaluation the probability of mass formation 6 months after cell injection.

SECONDARY OUTCOMES:
Hematoma | 1 month
  Evaluation the presence of hematoma 1 month after injection.
Muscle bulk | 6 months
  Evaluation the muscle bulk changes with sonography and MRI 6 months after transplantation.
CPK | 1month
  Evaluation the decrease of CPK 1 month after cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Department of Regenerative Medicine & Cell therapy center of Royan Institute; Mahdi Vahid Dastjerdi, MD, Study Director — Scientific Board of BouAli Hospital, Azad University; Leila Arab, MD, Principal Investigator — Department of Regenerative Medicine & cell therapy of Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org